CLINICAL TRIAL: NCT02804958
Title: Incheon-Bucheon Cohort of Patients Undergoing Primary Percutaneous Coronary Intervention for Acute ST-segment Elevation Myocardial Infarction
Brief Title: Incheon-Bucheon Cohort of Patients Undergoing Primary PCI for Acute STEMI
Status: Completed | Type: Observational
Sponsor: Gachon University Gil Medical Center (Other)
Collaborators: Soon Chun Hyang University (Other); Sejong General Hospital (Other); Inha University Hospital (Other)
Responsible Party: Principal Investigator, Woong Chol Kang, Professor, Gachon University Gil Medical Center
Other Study IDs: INTERSTELLAR
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Myocardial Infarction
Keywords: ST-segment elevation myocardial infarction; Primary percutaneous coronary intervention; Clinical outcomes
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- STEMI treated with primary PCI: Patients diagnosed with acute ST-segment elevation myocardial infarction and treated with primary percutaneous coronary intervention were consecutively registered.
  Interventions: Procedure: STEMI treated with primary PCI

INTERVENTIONS:
Procedure: STEMI treated with primary PCI — Primary percutaneous coronary intervention was performed according to the current standard guidelines. Coronary angiography was performed using standard techniques. The use of thrombectomy devices, intravascular ultrasound, intra-aortic balloon pump, and percutaneous cardiopulmonary support was up to the operator.

SUMMARY:
INcheon-Bucheon cohorT of patients undERgoing primary percutaneous coronary intervention for acute ST-ELevation myocardiaL infARction (INTERSTELLAR) registry is a retrospective, observational, 4-regional-hospital based registry reflecting current practices of management, risk factors, and clinical outcomes in patients with ST-segment elevation myocardial infarction undergoing primary percutaneous coronary intervention at cities of Incheon and Bucheon located in the mid-western part of the Korean peninsula between 2007 and 2014.

DETAILED DESCRIPTION:
INcheon-Bucheon cohorT of patients undERgoing primary percutaneous coronary intervention for acute ST-ELevation myocardiaL infARction (INTERSTELLAR) registry is a retrospective, observational, 4-regional-hospital based registry reflecting current practices of management, risk factors, and clinical outcomes in patients with ST-segment elevation myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention (PCI) at cities of Incheon and Bucheon located in the mid-western part of the Korean peninsula between 2007 and 2014. Diagnosis of acute STEMI was based on clinical data findings including typical symptoms, 12-lead electrocardiography, and blood test. Decisions regarding primary PCI were made by at least 2 attending cardiologists at the time of presentation.

Demographic data, cardiovascular risk factors, laboratory data and clinical follow-up data were collected. Baseline blood test was obtained and recorded as part of the routine care for patients who visited the emergency room for chest pain and in whom acute coronary syndrome was suspected. Standard medical management was provided by responsible physicians.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acute ST-segment elevation myocardial infarction
* Patients treated with primary percutaneous coronary intervention

Exclusion Criteria:

* Patients diagnosed with Non-ST-segment elevation acute coronary syndrome
* Patients treated with thrombolytic therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with acute ST-segment elevation myocardial infarction (STEMI) and treated with primary percutaneous coronary intervention (PCI) were consecutively registered. Diagnosis of acute STEMI was based on clinical data findings including typical symptoms, 12-lead electrocardiography, and blood test. Decisions regarding primary PCI were made by at least 2 attending cardiologists at the time of presentation.
Sampling Method: Probability Sample
Enrollment: 1537 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
MACCE | Within the 1 year
  Major adverse cardiac and cerebrovascular event (MACCE), defined as the composite of all-cause death, non-fatal myocardial infarction and non-fatal stroke

SECONDARY OUTCOMES:
All-cause death | Within the 1 year
Non-fatal myocardial infarction | Within the 1 year
Non-fatal stroke | Within the 1 year
Ischemic-driven revascularization | Within the 1 year
Admission for heart failure | Within the 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Woong Chol Kang, MD, Principal Investigator — Gachon University Gil Medical Center
Locations (4):
- South Korea (4):
  - Sejong General Hospital, Bucheon-si
  - Soon Chun Hyang University Bucheon Hospital, Bucheon-si
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon

IPD SHARING:
Plan to Share IPD: No